CLINICAL TRIAL: NCT05502601
Title: Impact of Non-surgical Periodontal Therapy in the Systemic and Clinical Conditions of Patients With Rheumatoid Arthritis: a 6-months Randomized Controlled Trial
Brief Title: Periodontal Therapy in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Universidad Científica del Sur (Other)
Responsible Party: Principal Investigator, Alex Nogueira Haas, Associate Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CientificaDelSur
Record Dates: First submitted 2022-04-01; First posted 2022-08-16 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Arthritis, Rheumatoid; Periodontitis
Keywords: C-reactive protein; Periodontal diseases; Periodontitis; Rheumatoid arthritis; Scaling and root planning
MeSH Terms: conditions — Arthritis, Rheumatoid; Periodontitis; Periodontal Diseases | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will be comprised by those who will not receive any specific oral care intervention. For ethical reasons, the control group will receive periodontal therapy at the Endo of the study (after 6 months). In those cases presenting periodontal disease progression in a single tooth, the patients will be treated and withdrawn from the study
- Non-surgical periodontal treatment (Active Comparator): Periodontal treatment will be performed with scaling and root planning (SRP).SRP will be performed under local anesthesia during a single, 2-hour, full-mouth ultrasonic and hand instrument debridement using curettes.
  Oral hygiene instructions (patient education and motivation to control plaque and calculus accumulation)
  Interventions: Procedure: Non-surgical periodontal treatment

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — SRP will be performed under local anesthesia during a single, 2-hour, full-mouth ultrasonic and hand instrument debridement using curettes.
  Oral hygiene instructions (to educate and motivate patients to control the accumulation of plaque and calculus)
  Other Names: Scaling and root planing
  Arms: Non-surgical periodontal treatment

SUMMARY:
Aim: A prospective randomized, controlled clinical trial comparing two groups of a cohort of Rheumatoid Arthritis (RA) patients with periodontal disease will be carried out to identify if the effect of non-surgical periodontal therapy is a predictor of remission/ low disease activity (LDA)-remission.

Methods: 42 patients with RA and periodontitis from the RA Almenara cohort will be included (ACR 1987 and or ACR/EULAR 2010 criteria with more than 16 years old at diagnosis); those with <6 teeth, current infections, cancer or oral precancerous lesions, diabetics, Sjogren's syndrome, use of antibiotics or drugs associated with dry mouth and dental surgery, will be excluded. Periodontal Disease was defined by the presence of periodontitis stage 3 or 4 with at least 2 non-adjacent teeth with insertion loss >=5mm, probing depth >=5mm and bleeding on probing according with the 2018 periodontitis diagnostic criteria.

Two RA patients groups will be follow up by monthly visits. Patients will be divided into two groups (intervention and no intervention treatment). PD treatment will be performed by a qualified periodontist. No intervention group will receive PD treatment after 6 month visit because ethical principles. Disease activity will be determined according with DAS 28index, Clinical Disease Activity Index (CDAI) and Simple Disease Activity Index (SDAI) scores, C-reactive protein (CRP), the erythrocyte sedimentation rate (ESR), and rheumatoid factor levels will be registered before and after PD treatment (baseline, 3 and 6 months visits), and the differences between the groups will be analyzed and compared. Periodontal parameters including probing depth (PD), clinical attachment loss, and sulcus bleeding index (SBI) will be correlated with the factor levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* Age ≥16 years at the time of diagnosis and who do not meet criteria of overlap with any other autoimmune disease.
* Presence of six or more permanent teeth in the mouth, excluding third molars.
* Presence of periodontitis stage 3 or 4 with at least 2 non-adjacent teeth with insertion loss >=5mm, probing depth >=5mm and bleeding on probing according to Tonetti et al.[35].
* Willingness to attend all visits for the duration of the study.

Exclusion Criteria:

* Patients with Sjogren's syndrome

  * - Severe ongoing systemic infection.
  * - Associated dental infection
  * - History of oral cavity cancer or precancerous lesion.
  * - Use of local or systemic antibiotics in the last 3 months (including tetracyclines or other medication that could change the periodontal evaluation in the investigator's opinion, such as heparin alendronate, antivitamin K).
  * - Medications that induce gingival hyperplasia (such as phenytoin, warfarin or cyclosporine).
  * - Pregnant or breastfeeding women
  * - Participation in another intervention study.
  * Patients with a history of PD treatment in the last 6 months or previous dental surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the Disease Activity Score with 28-joint counts (DAS 28) | Baseline, 3 and 6 months after treatment
  The DAS28 includes a 28-swollen joint count (28SJC), 28-tender joint count (28TJC), ESR, and a patient global assessment of disease activity (PtGA) or GH (General Health) assessment on a VAS. It may also be calculated using C-reactive protein (CRP) level instead of Westergren ESR the unabbreviated scale title: Disease Activity Score (28-joint counts) A score greater than 5.1 indicates active disease and less than 3.2 indicates well-controlled disease. A score of less of than 2.6 indicates remission
Changes in the Simplified disease activity index (SDAI) | Baseline, 3 and 6 months after treatment
  The SDAI includes a 28-swollen joint count (28SJC), 28-tender joint count (28TJC), patient global assessment of disease activity (PtGA) on a 10-cm visual analog scale (VAS), provider global assessment of disease activity (PrGA) on a 10-cm VAS, and C-reactive protein (CRP) level in mg/dl.
  The unabbreviated scale title: Simplified disease SDAI is calculated as follows: SDAI = SJC + TJC +PtGA + EGA (Evaluator Global disease Activity) + CRP.
  activity index The SDAI has range from 0 to 86. higher scores mean a worse outcome.
Changes in the Clinical disease activity index (CDAI) | Baseline, 3 and 6 months after treatment
  The CDAI includes a 28-swollen joint count (28SJC), 28-tender joint count (28TJC), patient global assessment of disease activity (PtGA) on a 10-cm visual analog scale (VAS), and provider global assessment of disease activity (PrGA) on a 10-cm VAS
  The unabbreviated scale title: Clinical disease activity index The CDAI has range from 0 to 76. higher scores mean a worse outcome.
Changes in Antibodies to cyclic citrullinated protein (anti-CCP) | Baseline, 3 and 6 months after treatment
  measurement of CCP (cyclic citrullinated peptide) antibodies in the blood
Changes in rheumatoid factor (RF) | Baseline, 3 and 6 months after treatment
  measurement of the amount of the RF antibody in the blood
Changes in erythrocyte sedimentation rate (ESR) | Baseline, 3 and 6 months after treatment
  measurement of the erythrocyte sedimentation rate in a test tube
C-reactive protein (CRP) | Baseline, 3 and 6 months after treatment
  measurement of the level of c-reactive protein (CRP) in your blood.

SECONDARY OUTCOMES:
Changes in Probing pocket depth (PPD) | Baseline, 3 and 6 months after treatment
  Measurement of pocket depth with periodontal probe in 6 sites per tooth
Changes in Clinical attachment level (CAL) | Baseline, 3 and 6 months after treatment
  Measurement from the cemento-enamel junction to the total probing depth in 6 sites per tooth
Changes in Bleeding on probing (BOP) | Baseline, 3 and 6 months after treatment
  Bleeding present or absent within 20 s after palpation in 6 sites per tooth
Changes in Plaque index (PI) | Baseline, 3 and 6 months after treatment
  Presence or absence of bacterial plaque in 6 sites per tooth

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Vergara, Principal Investigator — Universidad Cientifica del Sur
Locations (1):
- Universidad Cientifica del Sur, Lima, Peru

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cheng Z, Meade J, Mankia K, Emery P, Devine DA. Periodontal disease and periodontal bacteria as triggers for rheumatoid arthritis. Best Pract Res Clin Rheumatol. 2017 Feb;31(1):19-30. doi: 10.1016/j.berh.2017.08.001. Epub 2017 Sep 1. PMID 29221594
- [Background] Genco RJ, Sanz M. Clinical and public health implications of periodontal and systemic diseases: An overview. Periodontol 2000. 2020 Jun;83(1):7-13. doi: 10.1111/prd.12344. PMID 32385880
- [Background] Gabriel SE, Michaud K. Epidemiological studies in incidence, prevalence, mortality, and comorbidity of the rheumatic diseases. Arthritis Res Ther. 2009;11(3):229. doi: 10.1186/ar2669. Epub 2009 May 19. PMID 19519924
- [Background] Schneeberger EE, Citera G, Maldonado Cocco JA, Salcedo M, Chiardola F, Rosemffet MG, Marengo MF, Papasidero S, Chaparro Del Moral R, Rillo OL, Bellomio V, Lucero E, Spindler A, Berman A, Duartes Noe D, Barreira JC, Lazaro MA, Paira SO. Factors associated with disability in patients with rheumatoid arthritis. J Clin Rheumatol. 2010 Aug;16(5):215-8. doi: 10.1097/RHU.0b013e3181e92d25. PMID 20577095
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Zhao X, Liu Z, Shu D, Xiong Y, He M, Xu S, Si S, Guo B. Association of Periodontitis with Rheumatoid Arthritis and the Effect of Non-Surgical Periodontal Treatment on Disease Activity in Patients with Rheumatoid Arthritis. Med Sci Monit. 2018 Aug 20;24:5802-5810. doi: 10.12659/MSM.909117. PMID 30124222
- [Background] Ceccarelli F, Saccucci M, Di Carlo G, Lucchetti R, Pilloni A, Pranno N, Luzzi V, Valesini G, Polimeni A. Periodontitis and Rheumatoid Arthritis: The Same Inflammatory Mediators? Mediators Inflamm. 2019 May 5;2019:6034546. doi: 10.1155/2019/6034546. eCollection 2019. PMID 31191116
- [Background] Calderaro DC, Correa JD, Ferreira GA, Barbosa IG, Martins CC, Silva TA, Teixeira AL. Influence of periodontal treatment on rheumatoid arthritis: a systematic review and meta-analysis. Rev Bras Reumatol Engl Ed. 2017 May-Jun;57(3):238-244. doi: 10.1016/j.rbre.2016.11.011. Epub 2017 Jan 4. English, Portuguese. PMID 28535896
- [Background] Silvestre FJ, Silvestre-Rangil J, Bagan L, Bagan JV. Effect of nonsurgical periodontal treatment in patients with periodontitis and rheumatoid arthritis: A systematic review. Med Oral Patol Oral Cir Bucal. 2016 May 1;21(3):e349-54. doi: 10.4317/medoral.20974. PMID 26946202
- [Background] Sun J, Zheng Y, Bian X, Ge H, Wang J, Zhang Z. Non-surgical periodontal treatment improves rheumatoid arthritis disease activity: a meta-analysis. Clin Oral Investig. 2021 Aug;25(8):4975-4985. doi: 10.1007/s00784-021-03807-w. Epub 2021 Jan 29. PMID 33515120